CLINICAL TRIAL: NCT00001174
Title: Bipolar Genetics: A Collaborative Study
Brief Title: Evaluation of the Genetics of Bipolar Disorder
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 800083; 80-M-0083
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12-29

CONDITIONS: Bipolar Disorder
Keywords: Affective Disorder; Depression; Genetic Polymorphisms; Major Depression; Genome-Wide Scan; Natural History; Panic Disorder; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Depression; Depressive Disorder, Major; Panic Disorder

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy volunteers
- Patients: Patients with bipolar disorder

SUMMARY:
This study looks to identify genes that may affect a person's chances of developing bipolar disorder (BP) and related conditions....

DETAILED DESCRIPTION:
Study Description:

This project uses genetic mapping and whole exome sequencing methods to identify genetic markers and variations that contribute to the risk of bipolar disorder, an often severe, heritable condition affecting about one percent of the population. Individuals diagnosed with bipolar disorder are studied, along with their relatives. Phenotypic information obtained from clinical interviews and family history is correlated with genotypic information obtained from genetic marker and whole exome sequencing methods.

Objectives:

Primary Objective:

Identify genes involved in bipolar disorder and related conditions so that better methods of diagnosis, treatment, and prevention can be developed.

Secondary Objectives:

1. To identify genes that shape the clinical picture or influence response to treatment.
2. To replicate our findings in independent samples. Genome-wide genotyping, whole exome sequencing, demographic, and phenotype data will be requested under the usual dbGaP Data Access procedures and analyzed along with existing phenotypic and genetic data.
3. To analyze the clinical data, including but not limited to the diagnostic categories, in order to identify between-family differences which might identify genetically meaningful subgroups of families.
4. To submit coded phenotypes, genotypes, and DNA from informative families to a national archival database.
5. To establish a catalog of induced pluripotent stem cells suitable for functional genomic studies of neurons and glia in culture.

Endpoints:

Primary Endpoint:

The primary endpoint of this study is the identification of genes involved in risk for developing bipolar disorder.

Secondary Endpoints:

1. Pedigree structure, representing known relationships and reported mental health of first, second, and third-degree relatives
2. Dimensional data on mental health symptoms obtained from the Past History Schedule, Mood Disorders Questionnaire, and Symptom Checklist (SCL-90)
3. Cognitive data based on measures of executive function, working memory, attention, verbal memory, visuospatial reasoning, and affect recognition.
4. Lithium response data collected through the Retrospective Assessment of the Lithium Response (Alda) Scale
5. History of traumatic life events elicited with the Life Events Checklist for DSM-5 (LEC-5)
6. Genotype data obtained from SNP arrays or whole-exome sequencing
7. Skin biopsy or additional blood sample from selected participants
8. Induced pluripotent stem cells obtained from reprogramming of skin or blood cells.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Male or female, aged 18 years and over. Children are excluded for the following reasons: age at onset of BD is usually later than age 18, the diagnostic and assessment instruments we use are not validated in children.
3. In good general health as evidenced by medical history or diagnosed with or exhibiting symptoms of bipolar disorder or related conditions not attributable to substance abuse, or neurological disease; OR a 1st or 2nd degree relative of an enrolled participant. Related conditions are defined as those found more often among relatives of people with bipolar disorder or which have been shown to be genetically correlated with bipolar disorder through molecular genetic studies. These include major depression, schizophrenia, panic disorder, and attention deficit hyperactivity disorder.
4. Ability to safely provide a blood or saliva sample.
5. Ability of subject to understand and willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Active alcohol or substance abuse.
2. Subjects who suffer cognitive impairment and are unable to provide an accurate psychiatric history are excluded since much of the diagnostic information relies on selfreport and recall of past events.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community samples and clinical samples
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 1994-08-11 (Actual)

PRIMARY OUTCOMES:
Diagnosis of bipolar disorder or related mental illness by direct interview | Diagnosis is established primarily at the initial study visit. Participants who consent to recontact are re-evaluated when they or family informants report events that could lead to a revised diagnosis.
  Psychiatric diagnosis is based on systematic review of established signs and symptoms, using an instrument designed to elicit retrospective information of known reliability, supplemented with information from family informants, any medical records, and by dimensional symptom measures.

CONTACTS AND LOCATIONS:
Overall Officials: Francis J McMahon, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Amare AT, Thalamuthu A, Schubert KO, Fullerton JM, Ahmed M, Hartmann S, Papiol S, Heilbronner U, Degenhardt F, Tekola-Ayele F, Hou L, Hsu YH, Shekhtman T, Adli M, Akula N, Akiyama K, Ardau R, Arias B, Aubry JM, Hasler R, Richard-Lepouriel H, Perroud N, Backlund L, Bhattacharjee AK, Bellivier F, Benabarre A, Bengesser S, Biernacka JM, Birner A, Marie-Claire C, Cervantes P, Chen HC, Chillotti C, Cichon S, Cruceanu C, Czerski PM, Dalkner N, Del Zompo M, DePaulo JR, Etain B, Jamain S, Falkai P, Forstner AJ, Frisen L, Frye MA, Gard S, Garnham JS, Goes FS, Grigoroiu-Serbanescu M, Fallgatter AJ, Stegmaier S, Ethofer T, Biere S, Petrova K, Schuster C, Adorjan K, Budde M, Heilbronner M, Kalman JL, Kohshour MO, Reich-Erkelenz D, Schaupp SK, Schulte EC, Senner F, Vogl T, Anghelescu IG, Arolt V, Dannlowski U, Dietrich D, Figge C, Jager M, Lang FU, Juckel G, Konrad C, Reimer J, Schmauss M, Schmitt A, Spitzer C, von Hagen M, Wiltfang J, Zimmermann J, Andlauer TFM, Fischer A, Bermpohl F, Ritter P, Matura S, Gryaznova A, Falkenberg I, Yildiz C, Kircher T, Schmidt J, Koch M, Gade K, Trost S, Haussleiter IS, Lambert M, Rohenkohl AC, Kraft V, Grof P, Hashimoto R, Hauser J, Herms S, Hoffmann P, Jimenez E, Kahn JP, Kassem L, Kuo PH, Kato T, Kelsoe J, Kittel-Schneider S, Ferensztajn-Rochowiak E, Konig B, Kusumi I, Laje G, Landen M, Lavebratt C, Leboyer M, Leckband SG, Tortorella A, Manchia M, Martinsson L, McCarthy MJ, McElroy S, Colom F, Millischer V, Mitjans M, Mondimore FM, Monteleone P, Nievergelt CM, Nothen MM, Novak T, O'Donovan C, Ozaki N, Pfennig A, Pisanu C, Potash JB, Reif A, Reininghaus E, Rouleau GA, Rybakowski JK, Schalling M, Schofield PR, Schweizer BW, Severino G, Shilling PD, Shimoda K, Simhandl C, Slaney CM, Squassina A, Stamm T, Stopkova P, Maj M, Turecki G, Vieta E, Veeh J, Witt SH, Wright A, Zandi PP, Mitchell PB, Bauer M, Alda M, Rietschel M, McMahon FJ, Schulze TG, Clark SR, Baune BT. Association of polygenic score and the involvement of cholinergic and glutamatergic pathways with lithium treatment response in patients with bipolar disorder. Mol Psychiatry. 2023 Dec;28(12):5251-5261. doi: 10.1038/s41380-023-02149-1. Epub 2023 Jul 11. PMID 37433967
- [Derived] Amare AT, Schubert KO, Hou L, Clark SR, Papiol S, Cearns M, Heilbronner U, Degenhardt F, Tekola-Ayele F, Hsu YH, Shekhtman T, Adli M, Akula N, Akiyama K, Ardau R, Arias B, Aubry JM, Backlund L, Bhattacharjee AK, Bellivier F, Benabarre A, Bengesser S, Biernacka JM, Birner A, Brichant-Petitjean C, Cervantes P, Chen HC, Chillotti C, Cichon S, Cruceanu C, Czerski PM, Dalkner N, Dayer A, Del Zompo M, DePaulo JR, Etain B, Jamain S, Falkai P, Forstner AJ, Frisen L, Frye MA, Fullerton JM, Gard S, Garnham JS, Goes FS, Grigoroiu-Serbanescu M, Grof P, Hashimoto R, Hauser J, Herms S, Hoffmann P, Hofmann A, Jimenez E, Kahn JP, Kassem L, Kuo PH, Kato T, Kelsoe JR, Kittel-Schneider S, Kliwicki S, Konig B, Kusumi I, Laje G, Landen M, Lavebratt C, Leboyer M, Leckband SG, Tortorella A, Manchia M, Martinsson L, McCarthy MJ, McElroy SL, Colom F, Mitjans M, Mondimore FM, Monteleone P, Nievergelt CM, Nothen MM, Novak T, O'Donovan C, Ozaki N, Osby U, Pfennig A, Potash JB, Reif A; Major Depressive Disorder Working Group of the Psychiatric Genomics Consortium; Reininghaus E, Rouleau GA, Rybakowski JK, Schalling M, Schofield PR, Schweizer BW, Severino G, Shilling PD, Shimoda K, Simhandl C, Slaney CM, Squassina A, Stamm T, Stopkova P, Maj M, Turecki G, Vieta E, Veeh J, Witt SH, Wright A, Zandi PP, Mitchell PB, Bauer M, Alda M, Rietschel M, McMahon FJ, Schulze TG, Baune BT. Association of polygenic score for major depression with response to lithium in patients with bipolar disorder. Mol Psychiatry. 2021 Jun;26(6):2457-2470. doi: 10.1038/s41380-020-0689-5. Epub 2020 Mar 16. PMID 32203155
- [Derived] Pisanu C, Congiu D, Costa M, Chillotti C, Ardau R, Severino G, Angius A, Heilbronner U, Hou L, McMahon FJ, Schulze TG, Del Zompo M, Squassina A. Convergent analysis of genome-wide genotyping and transcriptomic data suggests association of zinc finger genes with lithium response in bipolar disorder. Am J Med Genet B Neuropsychiatr Genet. 2018 Oct;177(7):658-664. doi: 10.1002/ajmg.b.32663. Epub 2018 Oct 14. PMID 30318722
- [Derived] International Consortium on Lithium Genetics (ConLi+Gen); Amare AT, Schubert KO, Hou L, Clark SR, Papiol S, Heilbronner U, Degenhardt F, Tekola-Ayele F, Hsu YH, Shekhtman T, Adli M, Akula N, Akiyama K, Ardau R, Arias B, Aubry JM, Backlund L, Bhattacharjee AK, Bellivier F, Benabarre A, Bengesser S, Biernacka JM, Birner A, Brichant-Petitjean C, Cervantes P, Chen HC, Chillotti C, Cichon S, Cruceanu C, Czerski PM, Dalkner N, Dayer A, Del Zompo M, DePaulo JR, Etain B, Falkai P, Forstner AJ, Frisen L, Frye MA, Fullerton JM, Gard S, Garnham JS, Goes FS, Grigoroiu-Serbanescu M, Grof P, Hashimoto R, Hauser J, Herms S, Hoffmann P, Hofmann A, Jamain S, Jimenez E, Kahn JP, Kassem L, Kuo PH, Kato T, Kelsoe J, Kittel-Schneider S, Kliwicki S, Konig B, Kusumi I, Laje G, Landen M, Lavebratt C, Leboyer M, Leckband SG, Tortorella A, Manchia M, Martinsson L, McCarthy MJ, McElroy S, Colom F, Mitjans M, Mondimore FM, Monteleone P, Nievergelt CM, Nothen MM, Novak T, O'Donovan C, Ozaki N, Osby U, Pfennig A, Potash JB, Reif A, Reininghaus E, Rouleau GA, Rybakowski JK, Schalling M, Schofield PR, Schweizer BW, Severino G, Shilling PD, Shimoda K, Simhandl C, Slaney CM, Squassina A, Stamm T, Stopkova P, Maj M, Turecki G, Vieta E, Volkert J, Witt S, Wright A, Zandi PP, Mitchell PB, Bauer M, Alda M, Rietschel M, McMahon FJ, Schulze TG, Baune BT. Association of Polygenic Score for Schizophrenia and HLA Antigen and Inflammation Genes With Response to Lithium in Bipolar Affective Disorder: A Genome-Wide Association Study. JAMA Psychiatry. 2018 Jan 1;75(1):65-74. doi: 10.1001/jamapsychiatry.2017.3433. PMID 29121268
- [Derived] Hou L, Heilbronner U, Degenhardt F, Adli M, Akiyama K, Akula N, Ardau R, Arias B, Backlund L, Banzato CEM, Benabarre A, Bengesser S, Bhattacharjee AK, Biernacka JM, Birner A, Brichant-Petitjean C, Bui ET, Cervantes P, Chen GB, Chen HC, Chillotti C, Cichon S, Clark SR, Colom F, Cousins DA, Cruceanu C, Czerski PM, Dantas CR, Dayer A, Etain B, Falkai P, Forstner AJ, Frisen L, Fullerton JM, Gard S, Garnham JS, Goes FS, Grof P, Gruber O, Hashimoto R, Hauser J, Herms S, Hoffmann P, Hofmann A, Jamain S, Jimenez E, Kahn JP, Kassem L, Kittel-Schneider S, Kliwicki S, Konig B, Kusumi I, Lackner N, Laje G, Landen M, Lavebratt C, Leboyer M, Leckband SG, Jaramillo CAL, MacQueen G, Manchia M, Martinsson L, Mattheisen M, McCarthy MJ, McElroy SL, Mitjans M, Mondimore FM, Monteleone P, Nievergelt CM, Nothen MM, Osby U, Ozaki N, Perlis RH, Pfennig A, Reich-Erkelenz D, Rouleau GA, Schofield PR, Schubert KO, Schweizer BW, Seemuller F, Severino G, Shekhtman T, Shilling PD, Shimoda K, Simhandl C, Slaney CM, Smoller JW, Squassina A, Stamm T, Stopkova P, Tighe SK, Tortorella A, Turecki G, Volkert J, Witt S, Wright A, Young LT, Zandi PP, Potash JB, DePaulo JR, Bauer M, Reininghaus EZ, Novak T, Aubry JM, Maj M, Baune BT, Mitchell PB, Vieta E, Frye MA, Rybakowski JK, Kuo PH, Kato T, Grigoroiu-Serbanescu M, Reif A, Del Zompo M, Bellivier F, Schalling M, Wray NR, Kelsoe JR, Alda M, Rietschel M, McMahon FJ, Schulze TG. Genetic variants associated with response to lithium treatment in bipolar disorder: a genome-wide association study. Lancet. 2016 Mar 12;387(10023):1085-1093. doi: 10.1016/S0140-6736(16)00143-4. Epub 2016 Jan 22. PMID 26806518
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1980-M-0083.html